CLINICAL TRIAL: NCT04615299
Title: Battlefield Acupuncture and Its Use In Multimodal Perioperative Anesthesia Care
Acronym: BFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesiology WSU/DMC-NorthStar (Other)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 060117M1F(V)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Acupuncture, Ear
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: The treatment group (Group 1) will receive postoperative auricular battlefield acupuncture. The control group (Group 2) will receive sham (placebo) postoperative auricular battlefield acupuncture.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham acupuncture covers will be placed on control participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Auricular acupuncture (Active Comparator): Auricular (Battlefield) acupuncture needles will be utilized in the test arm, location of needles and stickers will be placed according to 5 VA approved BFA auricular acupuncture points associated with PONV, pain, and anxiety respectively
  Interventions: Device: Auricular acupuncture
- Sham acupuncture (Sham Comparator): The control arm will receive sham or placebo acupuncture via pressing of a blunt needle on the specified BFA locations and then application of adhesive stickers. In the control group simulating acupuncture, the needles will never enter the patients' skin and will give the impression to the patient that the procedure has taken place.
  Interventions: Device: Auricular acupuncture

INTERVENTIONS:
Device: Auricular acupuncture — Auricular or Battlefield acupuncture is an auricular therapy which has been in existence for centuries, with roots tied to Eastern Asian medicine.

SUMMARY:
The study hypothesis is that perioperative Auricular (battlefield) acupuncture for general surgery and urology cases undergoing general anesthesia will decrease opioid requirements, postoperative pain, the incidence of PONV, and the incidence of perioperative anxiety in comparison to simulated (placebo) perioperative battlefield acupuncture.

DETAILED DESCRIPTION:
INTRODUCTION:

Battlefield acupuncture is an auricular therapy that has been used for centuries, with roots tied to Eastern Asian medicine. Ease of application, low cost, and minimal side effects make battlefield acupuncture a perioperative modality that has been linked to decreased morbidity and mortality in patients undergoing surgical procedures and anesthesia (1). In the United States, there is pressure by the government and the medical community to decrease opioid use, especially in the perioperative time period. Opiate use due to postoperative pain, postoperative nausea and vomiting (PONV), perioperative anxiety have all been linked to an increased hospital stay, increased morbidity, and mortality, and ultimately higher healthcare costs (2). Anesthesia providers can be trained in the application of acupuncture in the perioperative time period. Through analysis of rates of postoperative opioid use, postoperative nausea and vomiting and perioperative anxiety, the efficacy, and utility of battlefield acupuncture will be realized as an effective adjunct to multimodal anesthesia care.

STUDY DESIGN AND METHODS:

This will be a prospective randomized study to compare auricular battlefield acupuncture to sham auricular battlefield acupuncture in patients undergoing general surgery and urology cases with general anesthesia. Participants in the study will be randomly assigned to either receive auricular battlefield acupuncture (treatment group) or simulated (placebo; control group) auricular battlefield acupuncture. Battlefield acupuncture needles will be utilized in the test arm and blunt needle pressing and covering with acupuncture stickers will be utilized in the control arm as a sham treatment. Location of needles and stickers will be placed according to 5 VA approved BFA auricular acupuncture points associated with PONV, pain, and anxiety respectively (Figure 1; 3). In both arms, the treatment ear will be covered after treatment so as to blind the patient. Both battlefield acupuncture and control groups will receive small band aids on the battlefield acupuncture needle sites. Both the evaluators for post procedure assessment along with the patient will be blinded in regards to what group they are in.

Inclusion Criteria:

1- Patients with an American Society of Anesthesiologists (ASA) Physical Status classification of 1 to 4 2 - Patients aged between 18 and 100 scheduled to undergo scheduled suitable inpatient/outpatient cases under anesthesia.

3 - Patients must be willing and fit to give written informed consent 4 - Inpatient stay required

Exclusion Criteria:

1. - Coagulopathies
2. - Patients with continuous epidural
3. - Uncooperative patient
4. - Psychiatric disorders and language deficiencies that may interfere with the assessment of pain
5. - Insufficient understanding of the pain scoring system.
6. - Outpatient stay

This study will be performed at the John D. Dingell VA Medical Center. Only a trained MD anesthesiologist will recruit patient in the preoperative period, where informed consent will be obtained. Computerized randomization will take place at the time the patient presents for surgery. Consent will be taken preoperatively.

Anesthetic Plan:

The anesthetic management will be general anesthesia with the provision of intravenous opioids intraoperatively and during recovery. Fentanyl will be the sole intra operative opioid. No other alterations of anesthetic management will take place pre or intra operatively. The battlefield acupuncture or sham battlefield acupuncture will be placed in the postoperative care unit (PACU).

Acupuncture Plan:

Typically acupuncture needles which are semi-permanent needles have the characteristics of remaining in the ear acupoints for up to 3-4 days before being pushed out toward to the surface by the previous flattened epidermis. The test arm (treatment group) will received actual acupuncture needles, while the control arm will received sham or placebo acupuncture via pressing of a blunt needle on the specified BFA locations and then application of adhesive stickers. In the control group simulating acupuncture, the needles will never enter the patients' skin and will give the impression to the patient that the procedure has taken place. The ear treated will be covered with a bandage via non-skin sensitive tape so as to blind the patient to which treatment group they are in.

Statistical Analysis:

An unpaired students-t-test procedure (two-sample assuming equal variances, two-tail significance p<0.05, 95% confidence interval) was performed to examine mean differences between the two study groups on all continuously scaled variables. A Repeated measures ANOVA will be used to measured differences between time for continuous variables at the 2 measured time points (1 hour and 24 hours). Assumptions of normality and/or homogeneity of variance will be checked and verified. Comparisons between study groups on proportional differences will be examined using a non-parametric Fisher's Exact Chi-square test, when applied to 2x2 tables. Statistical significance will be set at a p-value ≤0.05. All continuous data will be expressed as the mean with 95% upper and lower confidence intervals or Mean ± Standard deviation.

A binary outcome, superiority power analysis based on a rate of 33% reduction of opioid consumption in the auricular battlefield acupuncture group compared to controls (sham auricular battlefield acupuncture) concluded 72 participants (36 patients per group) would be necessary to achieve 80% power with a p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1- Patients with an American Society of Anesthesiologists (ASA) Physical Status classification of 1 to 4 2 - Patients aged between 18 and 100 scheduled to undergo scheduled suitable inpatient/outpatient cases under anesthesia.

3 - Patients must be willing and fit to give written informed consent 4 - Inpatient stay required

Exclusion Criteria:

1. - Coagulopathies
2. - Patients with continuous epidural
3. - Uncooperative patient
4. - Psychiatric disorders and language deficiencies that may interfere with the assessment of pain
5. - Insufficient understanding of the pain scoring system.
6. - Outpatient stay

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padmavathi Patel, MD, Principal Investigator — Wayne State University, John D. Dingell VA Medical Center
Locations (1):
- John D. Dingell VA Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Z, Dong H, Wang Q, Xiong L. Perioperative acupuncture modulation: more than anaesthesia. Br J Anaesth. 2015 Aug;115(2):183-93. doi: 10.1093/bja/aev227. PMID 26170347
- [Background] Fleckenstein J, Baeumler PI, Gurschler C, Weissenbacher T, Simang M, Annecke T, Geisenberger T, Irnich D. Acupuncture for post anaesthetic recovery and postoperative pain: study protocol for a randomised controlled trial. Trials. 2014 Jul 21;15:292. doi: 10.1186/1745-6215-15-292. PMID 25047046

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 23 | 22 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 33 | 34 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (NIH/OMB): Black or African American | 14 | 19 | 33
  Race (NIH/OMB): White | 18 | 12 | 30
  Race (NIH/OMB): Other or Not Reported | 4 | 5 | 9
Body Mass Index [Mean (Standard Deviation); unit: Kg/(m^2)] | 30.1 (6.1) | 28.8 (5.9) | 29.5 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Consumption
Description: Patient opioid consumption in the 24 hrs post surgery
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalent
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
Morphine Milligram Equivalent | 18.3 (12.2) | 38.6 (15.9)

2. Primary Outcome: Pain Score Visual Analog Scale (VAS) 6 Hours Post Surgery
Description: Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
units on a scale | 4.3 (1.9) | 6.8 (1.9)

3. Primary Outcome: Pain Score Visual Analog Scale (VAS) 12 Hours Post Surgery
Description: Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
score on a scale | 3.6 (1.7) | 5.6 (1.6)

4. Primary Outcome: Pain Score Visual Analog Scale (VAS) 18 Hours Post Surgery
Description: Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
score on a scale | 3.1 (1.5) | 5.6 (1.6)

5. Primary Outcome: Pain Score Visual Analog Scale (VAS) 24 Hours Post Surgery
Description: Pain score on an 11-point (0 - no pain to 10 - worst imaginable pain) Visual Analog Scale (VAS) at rest
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
score on a scale | 2.3 (1.4) | 5.3 (2.0)

6. Secondary Outcome: Occurrence of Postoperative Vomiting
Description: Any patient incidence of vomiting within the 24 hour period post-surgery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
Participants | 0 | 11

7. Secondary Outcome: Occurrence of Postoperative Nausea
Description: Any reported patient incidence of nausea within the 24 hour period post-surgery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
Participants | 1 | 13

8. Secondary Outcome: Occurrence of Postoperative Anxiety
Description: Any patient incidence of postoperative anxiety within the 24 hr period post-surgery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
Participants | 4 | 5

9. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction of analgesia scoring from a range of (0% -very unsatisfied to 100% -extremely satisfied)
Time Frame: 24 hours
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
score on a scale | 8 [4 to 8] | 6 [2 to 8]

10. Secondary Outcome: Occurrence of Any Adverse Reactions
Description: Any occurrence of acupuncture site infection, acupuncture site bleeding, allergic reaction to acupuncture needles, or scar tissue formation at site of acupuncture needle within the 24-hr period post-surgery
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 36 | 36
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours post-surgery
Description: Adverse events were defined as any of the following reported within 24 hours following surgery including acupuncture site infection, acupuncture site bleeding, allergic reaction to acupuncture needles, and scar tissue formation at the site of acupuncture placement.
Arm/Group | Auricular Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04615299/Prot_SAP_ICF_001.pdf